CLINICAL TRIAL: NCT00435383
Title: Oxygen Saturation During Transfer From Operating Room to Post Anesthesia Care Unit After Current Anesthesia Care
Brief Title: Comparing Oxygen Saturation in Post Anesthesia Care Unit After Different Methods of Pain Relief
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Samia Khalil, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-02-220
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Cryptorchidism
Keywords: Caudal Block; Oxygen Saturation; Uni or Bilateral Orchidopexy
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational: Group 1 received a presurgical caudal block and group 2 received a intravenous narcotics.

SUMMARY:
To determine the which method of pain relief is better after current anesthesia care.

DETAILED DESCRIPTION:
We hypothesized that in children, the current anesthesia care (combined light general anesthesia and caudal analgesia) may decrease incidence of intra and or postoperative de-saturation( SaO2 < %95), the need of oxygen during child's transport to the PACU and during his stay in the recovery room, compared with children who receive intravenous narcotics for intra and postoperative pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* ASA physical status 1 or 2
* 1-6 yr old
* Scheduled for elective uni or bilateral orchidopexy

Exclusion Criteria:

* Children with compromised pulmonary, cardiac, neurological, hematological, renal condition, with history of prematurely or are obese will be excluded.

Ages: 1 Year to 6 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children scheduled for elective uni or bilateral orchidopexy.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2003-03; Primary Completion 2007-02 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samia Khalil, M.D., Principal Investigator — University of Texas, Houston, Texas
Locations (1):
- University of Texas,Anesthesiology Department, Houston, Texas, United States